CLINICAL TRIAL: NCT06269354
Title: Multi-center Study on Comprehensive Diagnosis and Treatment of Lower Limb Bone Defect Based on Three-dimensional Printing Technology
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20231121-71479
Record Dates: First submitted 2023-12-18; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: Bone Defects
Keywords: 3D printing technology; bone defects; clinical effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Traumatic bone defect in lower limb: Traumatic bone defect in lower limb
  Interventions: Device: 3D printed prostheses
- Infective lower limb bone defect: Infective lower limb bone defect
  Interventions: Device: 3D printed prostheses
- Neoplastic bone defect in lower limb: Neoplastic bone defect in lower limb
  Interventions: Device: 3D printed prostheses

INTERVENTIONS:
Device: 3D printed prostheses — 3D printed prostheses

SUMMARY:
The clinical diagnosis and treatment of lower limb bone defect is a difficult problem in orthopedics. The traditional treatment has the shortcomings of long treatment period, no weight bearing in the early stage of the limb, weak mechanical strength, many complications, and difficulty in repairing deformed and large segment bone defects around the joint. The Orthopedics Department of Peking University Third Hospital, the lead unit of this study, developed the TCBridge system based on three-dimensional (3D) printing technology in the early stage, which is the first approved 3D printing lower limb long bone defect repair system in China. The system can achieve personalized and accurate repair of lower limb bone defects, and ensure patients to carry out limb weight and functional exercise safely in the early stage after surgery. On this basis, this study will establish a multi-center clinical case cohort to achieve accurate comprehensive diagnosis and treatment of lower limb bone defects, benefiting patients and contributing to society.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with traumatic lower limb bone defect;
2. Infected lower limb bone defect patients;
3. Patients with neoplastic lower limb bone defect;
4. The above reasons caused bone defects of more than 5CM
5. at least 18 years of age;
6. Sign an informed agreement and join the study cohort voluntarily.

Exclusion Criteria:

1. Patients who do not agree to the use of 3D printed microporous titanium alloy prostheses;
2. Patients who cannot tolerate surgery;
3. the subjects cannot comply with the follow-up or affect the scientific and integrity of the study;
4. Other patients who were not suitable for inclusion as assessed by clinicians.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower limb defects
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of implant stability, new bone growth- limb length | post-operative 1.3.6.12.24.36 months
  X-ray X、CT images
Evaluation of bone healing | post-operative 3.6.12.24.36 months
  computed tomography (CT)

SECONDARY OUTCOMES:
Pain assessment | post-operative 1.3.6.12.24.36 months
  Visual Analog Score (VAS), total score is 10, "0" represents no pain, "10" represents the most unbearable pain
Evaluation of life quality and health status. | post-operative 1.3.6.12.24.36 months
  36-item short form survery (SF-36) questionnaire, it includes 8 itmem, namely physical functioning, vitality, bodily pain, general health, social functioning, role physical, role emotional, mental health. The maximum score of each item is 100, higher score represents better result.
Evaluation of knee function | post-operative 1.3.6.12.24.36 months
  hospital for special surgery (HSS) score. The maximum score of HSS is 100, higher score represents better result.
Evaluation of hip function | post-operative 1.3.6.12.24.36 months
  Harris score, The maximum score of Harris score is 100, higher score represents better result.
Evaluation of ankle function | post-operative 1.3.6.12.24.36 months
  American Orthopaedic Foot & Ankle Society (AOFAS) score，The maximum score of AOFAS score is 100, higher score represents better result.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No